CLINICAL TRIAL: NCT04110444
Title: Sildenafil Citrate Added to Low Molecular Weight Heparin and Low Dose Aspirin to Improve Uteroplacental Perfusion in High-risk Pregnancy
Brief Title: Sildenafil Citrate Added to Low Molecular Weight Heparin and Low Dose Aspirin in High-risk Pregnancy
Status: Withdrawn | Type: Observational
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Sahar MY Elbaradie, associate Professor, Fayoum University Hospital
Other Study IDs: SMElbaradie
Record Dates: First submitted 2019-09-26; First posted 2019-10-01 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: High Risk Pregnancy
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sildenafile group A: received sildenafil citrate orally 20mg every 8 hours based on previous studies18,21 (Respatio tablet, pharma Egypt group) in addition to low molecular weight heparin daily according to the bodyweight at the booking visit (Clexane 20,40,60 mg, Sanofi eventis company) plus small dose of aspirin 75 mg (Aspocid 75mg tablet, CID pharmaceutical) once daily
  Interventions: Drug: Sildenafil
- control group B: received low molecular weight heparin as subcutaneous injection once daily plus low dose aspirin 75mg orally once daily in addition to placebo three times daily prepared by a local pharmacy from a domestic manufacturer

INTERVENTIONS:
Drug: Sildenafil — oral sildenafil t.d.s for high-risk pregnancies
  Groups: sildenafile group A

SUMMARY:
Anticoagulant therapy is indicated during pregnancy for the prevention and treatment of venous thromboembolism, systemic embolism in patients with mechanical heart valves and, in combination with aspirin, for the prevention of recurrent pregnancy loss in women with antiphospholipid antibodies Sildenafil citrate increases uterine blood flow and potentiates estrogen-induced vasodilatation. Intravaginal administration of Sildenafil in the success of in vitro fertilization describes no deleterious effects on mother and fetus

DETAILED DESCRIPTION:
Pregnancy is considered an acquired hypercoagulable state due to increased concentration of coagulation factors, decreased levels of anticoagulants and decreased fibrinolytic capacity. Adverse pregnancy outcomes affect up to 15% of gestations and are the major cause of maternal and fetal morbidity and mortality. A poor perinatal outcome is expected in pregnancies with high vascular resistance in uterine circulation, but the pregnancies in which the resistance values are normalized in the later trimesters have a significantly better outcome.

For the prevention of fetal growth restriction, a recent large-study level meta-analysis and individual patient data meta-analysis confirm that aspirin modestly reduces small-for-gestational-age pregnancy in women at high risk (relative risk, 0.90, 95% confidence interval, 0.81-1.00) and that a dose of ≥100 mg should be recommended and to start at or before 16 weeks of gestation. Moreover, in vitro and in vivo studies suggest that low-molecular-weight heparin may prevent fetal growth restriction; however, evidence from randomized control trials is inconsistent.

In a normal pregnancy, the trophoblast produces nitric oxide (NO) which plays an important role in vasodilatation in the fetoplacental circulation to improve oxygen and nutritional supply to the fetus (9,10). Nitric oxide relaxes arterial and venous smooth muscle potently and might inhibit platelet aggregation and adhesion. Moreover, increased circulating phosphodiesterase (PDE) activity is suspected in women with preeclampsia. In pregnancies with fetal growth restriction and without preeclampsia, a reversible increased myometrial arterial tone by phosphodiesterase inhibition has been reported in vitro.

Phosphodiesterase type 5 inhibitors that potentiate nitric oxide availability such as sildenafil citrate have been extensively researched both in preclinical and clinical studies; Sildenafil citrate is a selective inhibitor of cyclic guanosine monophosphate (cGMP)-specific phosphodiesterase (PDE)-5 leading to cyclic guanosine monophosphate (cGMP) accumulation and enhances the relaxation elicited by exogenous and neural-released nitric oxide in corpus cavernous. Sildenafil citrate increases uterine blood flow and potentiates estrogen-induced vasodilatation. Intravaginal administration of Sildenafil in the success of in vitro fertilization describes no deleterious effects on mother and fetus. The Natural Killer Cells activity and endometrial thickness were significantly changed after vaginal Sildenafil therapy so it might be an interesting therapeutic option before conception in women with recurrent reproductive failure.

Reduced flow / increased resistance in uterine and umbilical arteries, indicative of reduced uteroplacental flow in pregnancies with fetal growth restriction, has been documented by non-invasive Doppler ultrasound velocimetry.

ELIGIBILITY:
Inclusion Criteria:

* high-risk pregnant women (women with current preeclampsia, IUGR and oligohydramnios)
* gestational age 28-37 weeks
* no major medical illness contraindicating sildenafil use (cardiovascular disease, sickle cell anaemia, retinopathy, hearing loss, liver diseases)
* willingness to sign informed consent for study randomization

Exclusion Criteria:

* gestational age less than 28 weeks
* refusal of Doppler studies or sildenafil use
* contraindication or allergy to sildenafil
* those who can't present for monitoring visits or follow medication instructions
* those with major medical illness including cardiovascular disease and diabetes mellitus
* multiple pregnancies
* suspected chromosomal or fetal congenital anomalies (documented by level II ultrasound examination)
* users of any vasodilator agents
* those who had maternal or fetal emergencies necessitating delivery at time of recruitment in the study or with diastolic blood pressure more than 110 mmHg
* BMI is more than 34 that would impede accurate measurement of fetal biometry and Doppler parameters

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: high-risk pregnant women of gestational age 28-37 weeks women with current preeclampsia, IUGR and oligohydramnios
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
change in abdominal circumference and estimated fetal weight after 2 weeks of therapy | two weeks
  ultrasound assessment of fetal growth

SECONDARY OUTCOMES:
amniotic fluid index 5-15 cm with minimum increase of 2 cm | two weeks
  ultrasound assessment of amniotic fluid

CONTACTS AND LOCATIONS:
Locations (1):
- sahar M.Y elbaradie, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided